CLINICAL TRIAL: NCT03383432
Title: Ultrasound-guided Approach Versus Uterine Sound-sparing Approach for Intrauterine Device Insertion a Randomized Clinical Trial
Brief Title: Intrauterine Device Insertion: a Step for High Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUD-TAUSSA
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Intrauterine Device
MeSH Terms: interventions — Intrauterine Devices; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-abdominal ultrasound intrauterine device group. (Other): Those will be subjected to intrauterine device insertion under trans-abdominal ultrasound guidance. In this method the participant will be asked to have a full bladder. Full bladder helps to displace the bowel out of the pelvis and acts as an acoustic window for high frequency sound waves and to straighten the angle between the uterine body and cervix in anteverted uterus, performing the function of the tenaculum. Then, then ultrasound will be done and the intrauterine device will be introduced vaginally under ultrasound vision.
  Interventions: Device: Intrauterine device; Radiation: Ultrasound
- Uterine Sounding Sparing intrauterine device group (Other): The sonographer performs ultrasound using transvaginal probe to evaluate the uterine position and the endometrial length in the sagittal view of the uterus. The intrauterine device was inserted directly into the uterine cavity without using uterine sounding.
  Interventions: Device: Intrauterine device; Procedure: uterine sounding sparing technique

INTERVENTIONS:
Device: Intrauterine device — Copper T 380 A
Radiation: Ultrasound — Transabdominal ultrasound
  Arms: Trans-abdominal ultrasound intrauterine device group.
Procedure: uterine sounding sparing technique — we will insert intrauterine device without using the uterine sound and we will replace this step by ultrasound before insertion
  Arms: Uterine Sounding Sparing intrauterine device group

SUMMARY:
The intrauterine device is a safe, reliable and long-acting reversible contraceptive method. Instrumentation of lower genital mucosa during intrauterine device application provokes pain because it is highly sensitive to touch. Fear of pain associated with intrauterine device insertion is considered a barrier to use this contraception method.

The classic insertion instructions recommend performing bimanual examination and uterine sounding prior to intrauterine device insertion in order to confirm proper determination of uterine size and position. The pain during intrauterine device insertion could be due to cervical grasping by the tenaculum, traction on the cervical canal, stretching of the internal os by the uterine sound or the intrauterine device inserter, and lastly by irritation of the endometrial lining by the intrauterine device.

Many studies investigated the use of various analgesics in different doses and routes of administration and found out that it has a significant impact on relieving of associated pain Some technical modifications have been emerged in trial to decrease pain during intrauterine device insertion. One of them is trans-abdominal ultrasound guided intrauterine device insertion which the participant with a full bladder is subjected to intrauterine device insertion under ultrasonographic guide without using tenaculum. This method effectively decreased the pain and time of intrauterine device insertion.

A recent method named "Uterine Sounding Sparing Approach" has been reported very recently in literature by Ali et al., 2017. In this method; the sonographer performs T transvaginal ultrasound to evaluate the uterine position and the endometrial length in the sagittal view of the uterus. The intrauterine device was inserted directly into the uterine cavity without using uterine sounding.

In spite of less pain reported by trans-abdominal ultrasound guided intrauterine device insertion (no vulsellum was used), this methods also have some drawbacks, firstly; the full bladder may displace the cervix upward making the intrauterine device application not quite easy and secondly; this method needs two investigators which may distress the women who wondering about this. These two drawbacks may decrease patient's and physician's satisfaction. The uterine sounding sparing approach lacks these two drawbacks which make it more satisfying.

From above evidence, there is a strong need to compare the satisfaction rate between the two mentioned approaches in trial to answer this question. Up to our knowledge; no randomized trial has been conducted or registered to compare the satisfaction rate between two above approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-49 years
2. Nonpregnant
3. Women did not receive any analgesics or misoprostol in the 24 hours prior to insertion.

Exclusion Criteria:

1. Women with any uterine abnormalities such as congenital anomalies, endometrial lesions, fibroids
2. Allergy to Copper.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Level of satisfaction of patients in both groups (satisfaction score) | 5 minutes after intrauterine device insertion
  Measured by visual analogue like scale from 0 to 10

SECONDARY OUTCOMES:
Level of reported pain (visual analogue scale ) | 5 minutes after intrauterine device insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided